CLINICAL TRIAL: NCT06336291
Title: A Dose Optimization Study for L19TNF in Combination With Lomustine in Patients With Glioblastoma at Progression or Recurrence
Brief Title: A Study With L19TNF in Combination With Lomustine in Patients With Glioblastoma at Progression or Recurrence
Acronym: GLIOSTELLA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFLOM-01/23
Record Dates: First submitted 2024-03-04; First posted 2024-03-28 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma
Keywords: L19TNF; Glioblastoma at progression
MeSH Terms: conditions — Glioblastoma | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm A (Experimental): Patients will be treated with L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26 and Lomustine on Day 1 (in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles.
  Interventions: Drug: L19TNF; Drug: Lomustine
- Arm B (Experimental): Patients will be treated with on Days 1, 3 and 5, and on Days 22, 24 and 26 and Lomustine on Day 1 (in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles
  Interventions: Drug: L19TNF; Drug: Lomustine
- Arm C (Experimental): Patients will be treated with L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26 and Lomustine on Day 1 (in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles.
  Interventions: Drug: L19TNF; Drug: Lomustine
- Arm D (Experimental): Patients will be treated with L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26 and Lomustine on Day 1 (in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles.
  Interventions: Drug: L19TNF; Drug: Lomustine
- Arm E (Experimental): Patients will be treated with L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26 and Lomustine on Day 1 (in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles.
  Interventions: Drug: L19TNF; Drug: Lomustine
- Arm F (Experimental): Patients will be treated with L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26 and Lomustine on Day 1 (in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles.
  Interventions: Drug: L19TNF; Drug: Lomustine

INTERVENTIONS:
Drug: L19TNF — 7 μg/kg
  Other Names: onfekafusp alfa
  Arms: Arm A; Arm B
Drug: L19TNF — 10 μg/kg
  Other Names: onfekafusp alfa
  Arms: Arm C; Arm D
Drug: L19TNF — 13 μg/kg
  Other Names: onfekafusp alfa
  Arms: Arm E; Arm F
Drug: Lomustine — 90 mg/m2
  Arms: Arm A; Arm C; Arm E
Drug: Lomustine — 110 mg/m2
  Arms: Arm B; Arm D; Arm F

SUMMARY:
The trial aims to collect safety, efficacy, exposure, dose- response, pharmacokinetic and pharmacodynamic information of the combination of L19TNF and lomustine at different dose levels in patients with Glioblastoma at progression or recurrence

DETAILED DESCRIPTION:
The present study is a randomized, open-label, non-controlled phase II study in patients with glioblastoma at any progression/recurrence (first and later).

Overall, 90 subjects will be enrolled and parallel assigned in a 1:1 fashion to one of six treatment arms (from A to F) of 15 patients each.

Each arm has a different combination of L19TNF (7 μg/kg or 10 μg/kg or 13 μg/kg) and lomustine at different dose levels (90 or 110 mg/m2).

Treatment is based on a 42-day cycle for up to a maximum of 6 cycles.

This is an open-label study, so there is no blinding.

Patients who successfully complete the screening evaluations and are eligible for participation in the study will be enrolled and randomly assigned (1:1:1:1:1:1) to either of the six parallel treatment arms.

To maintain an appropriate balance between the six treatment arms and avoid undesired confounding effect of different factors, patients will be randomized in accordance with the following strata:

* MGMT status
* Steroid administration
* Previous systemic therapy treatment for progression

A randomization list will be prepared for each stratum using permuted block, the block sizes will be chosen randomly from different, pre-specified sizes with an equal treatment allocation ratio. The labels for the arms are assigned randomly within each block (fixed seed). The obtained final list is sorted by block together with the progressive enrollment number for the patients.

The primary objective of this study is to select the optimal regimen of L19TNF in combination with lomustine, that maximizes effects on clinical parameters and minimizes the probability of moderate to severe adverse events, among six (three L19TNF doses x two lomustine doses) combination schedules for the treatment of patient with progressing or recurrent glioblastoma.

Primary endpoints include Safety (Incidence of adverse Events (AEs), Serious Adverse Events (SAEs) and Drug-Induced Liver Injury (DILI), standard laboratory assessments, ECG, ECHO and physical examination according to CTCAE v.5.0) and Efficacy (Survival rate at 12 months).

The secondary objective of this study is to further evaluate safety, efficacy, exposure, dose-response, pharmacokinetic and pharmacodynamic information of the combination of L19TNF and lomustine at different dose levels to determine the best dose regimen for further studies.

During the conduct of the study the safety information collected will be routinely reviewed by the Data and Safety Monitoring Board (DSMB) in order to identify possible safety concerns.

If the probability in a treatment arm that the development of unacceptable toxicity rate exceeds 33 % is equal or higher than 80%, the recruitment to this treatment arm will be interrupted and the DSMB will be informed to assess the events and relationship to the study treatment. The DSMB may then recommend to re-start recruitment again for the treatment arm or permanently suspend it.

In case of a treatment-related death, recruitment will be suspended for all treatment arms until the Data and Safety Monitoring Board (DSMB) has reviewed the event and recommended to restart

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18.
2. Patients with histologically confirmed glioblastoma per 2021 WHO classification progression according to RANO criteria.
3. For operated patients, the histological report must document glioblastoma recurrence and a new MRI will need to be done at 3-5 weeks after surgery (directly before study treatment start). Study treatment will need to start minimum 4 weeks after surgery.
4. MGMT promotor status known.
5. Karnofsky Performance Status (KPS) ≥ 60%.
6. Documented negative test for HIV-HBV-HCV. For HBV serology, the determination of HbsAg and anti-HbcAg Ab is required. In patients with serology documenting previous exposure to HBV, negative serum HBV-DNA is required (HBV-DNA is not required for patients with documented vaccination report). For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
7. Female patients: female patients must be either documented not Women Of Childbearing Potential (WOCBP)* or must have a negative pregnancy test within 14 days of starting treatment.

   Additionally WOCBP must agree to use, from the screening to 6 months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.
8. Male patients: male subjects able to father children must agree to use two acceptable methods of contraception throughout the study and until 6 months after last study drug administration (e.g. condom with spermicidal gel). Double-barrier contraception is required.
9. Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
10. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

    * Women of childbearing potential (WOCBP) are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).

Exclusion Criteria:

1. Inability to undergo contrast-enhanced MRI.
2. Anti-cancer treatment with radiation therapy, chemotherapy, targeted therapies, immunotherapy, hormones, tumor treating fields or other antitumor therapies within 4 weeks prior to study treatment start.
3. Subjects who participated in an investigational drug or device study within 4 weeks prior to study treatment start.
4. Grade ≥ 4 myelotoxicity with previous treatment of alkylating agents (e.g., TMZ, CCNU).
5. Previous treatment with Bevacizumab.
6. Previous treatment with L19TNF.
7. Previous treatment in the PH-L19TNFCCNU-02/20 study.
8. Known history of allergy to TNF, any excipient in the study medication or any other intravenously administered human proteins/peptides/antibodies.
9. Absolute neutrophil count (ANC) < 1.5 x 10^9/L; platelets < 100 x 10^9/L or hemoglobin (Hb) < 9.0 g/dl.
10. Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min/1.73m2 or for patients older than 65 years without albuminuria or proteinuria, creatinine clearance < 45 mL/min/1.73m2.
11. Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN or total bilirubin ≥ 1.5 x ULN).
12. INR > 1.5 ULN.
13. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
14. Active or history of autoimmune disease that might deteriorate when receiving an immune-stimulatory agent, in the judgement of the investigator.
15. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
16. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
17. Clinically significant cardiac arrhythmias or requiring permanent medication.
18. LVEF <55% or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator. Patients with a marked prolongation of QT/QTc interval (e.g., repeated demonstration of QTc >470 milliseconds using Fredricia's QT correction formula) are excluded.
19. Uncontrolled hypertension.
20. Known arterial aneurism at high risk of rupture.
21. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification)
22. Anxiety ≥ CTCAE Grade 3.
23. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
24. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 3 weeks of administration of study treatment.
25. Known active or latent tuberculosis (TB).
26. Pregnancy or breast feeding.
27. Requirement of chronic administration of high dose corticosteroids or other immunosuppressant drugs. Subjects must have been either off corticosteroids, or on a stable or decreasing dose ≤ 4 mg daily dexamethasone (or equivalent) for 7 days prior to start of treatment. Limited or occasional use of corticosteroids to treat or prevent acute adverse reactions is not considered an exclusion criterion.
28. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
29. Concurrent malignancies unless the patient has been disease-free without intervention for at least 2 years.
30. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
31. Serious, non-healing wound, ulcer, or bone fracture.
32. Deep vein thrombosis, pulmonary embolism or other acute vascular events within 6 months.
33. Anticoagulation therapy with P2Y12 antagonists (e.g., clopidogrel, ticagrelor) and vitamin K antagonists (e.g., phenprocoumon, warfarin).
34. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
35. Any recent live vaccination within 4 weeks prior to treatment or plan to receive live vaccination during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From the screening, throughout the study, until demonstration of confirmed disease progression, treatment begins with another anti-cancer agent or surgery, or for a minimum of 12 months
  Occurence of AEs according to CTCAE v.5.0
Serious Adverse Events | From the screening, throughout the study, until demonstration of confirmed disease progression, treatment begins with another anti-cancer agent or surgery, or for a minimum of 12 months
  Occurence of SAEs according to CTCAE v.5.0
Unacceptable Toxicity | From the start of treatment up to 3 months
  Occurence of Unacceptable Toxicity according to CTCAE v.5.0
DILI assessment | From the screening, throughout the study, until demonstration of confirmed disease progression, treatment begins with another anti-cancer agent or surgery, or for a minimum of 12 months
  Occurence of DILI according to CTCAE v.5.0
Survival | From enrollment to death from any cause, for a minimum of 12 months
  Survival rate at 12 months

SECONDARY OUTCOMES:
Overall Survival | From enrollment to death from any cause, for a minimum of 12 months
Progression Free Survival | From enrollment to the date of progression or death from any cause, whichever came first, for a minimum of 12 months
Objective Response Rate | From enrollment to death from any cause, for a minimum of 12 months
  The rate of patients achieving Complete Response (CR) or Partial Response (PR) defined according to RANO criteria
Disease Control Rate | From enrollment to death from any cause, for a minimum of 12 months
  The rate of patients achieving complete (CR), partial (PR) and stable response (SD)
Duration of Response | From enrollment to the date of progression or death from any cause, whichever came first, for a minimum of 12 months
Time to reach maximum drug concentration [Tmax] | From the start of treatment up to 9 months
  Pharmacokinetics assessment of L19TNF through blood sampling
Terminal half-life [t1/2] | From the start of treatment up to 9 months
  Pharmacokinetics assessment of L19TNF through blood sampling
Area under the drug concentration-time curve, extrapolated to infinity [AUC] | From the start of treatment up to 9 months
  Pharmacokinetics assessment of L19TNF through blood sampling
Maximum drug concentration [Cmax] | From the start of treatment up to 9 months
  Pharmacokinetics assessment of L19TNF through blood sampling
Human anti-fusion protein antibodies (HAFA) levels against L19TNF | From the start of treatment to the date of progression or death for any cause, whichever come first
  Determination of the formation of Human Anti-Fusion protein Antibodies (HAFA) against L19TNF

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Virginia (UVA), Charlottesville, Virginia